CLINICAL TRIAL: NCT03680924
Title: Access to Resources for Patients With PTEN Hamartoma Tumor Syndrome
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DSC 7907
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-02

CONDITIONS: PTEN Gene Mutation
Keywords: PTEN; phosphatase and tensin homology mutation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to gain a better understanding of access to clinical and research resources for families of children affected with a phosphatase and tensin homology (PTEN) mutation. Ultimately, the researchers hope to be able to use this information to develop a standard of care for affected individuals and their family members. Family members/legal guardians of an individual with a PTEN mutation enrolled in the Rare Diseases Clinical Research Network (RDCRN) Contact Registry will be invited via email to participate in this study.

DETAILED DESCRIPTION:
The purpose of this study is to investigate access to clinical care and clinical research for patients with PTEN hamartoma tumor syndrome. This research will entail an anonymous online survey sent to families/caretakers of affected children. The survey will inquire: (1) basic clinical information about the child, such as diagnoses (both genetic and neurodevelopmental), level of functioning (estimated IQ) (2) clinical specialists that the child sees or needs to see (3) how families learn about clinical trials/research relevant to their child (4) basic demographics about the parent/caretaker completing the survey.

Specifically, this survey will collect information pertaining to:

* Number of affected children in household
* PTEN mutation type of affected children
* Age and gender of affected children
* Age, neurodevelopmental disorders, medical problems, IQ, and access to clinical care (specialists currently being seen, specialists not able to see and why) of most affected child
* Research methods and mediums for disorder-specific treatment options for affected children
* Reasons behind not participating in clinical research options
* Facts (gender, age, if PTEN mutation carrier, work status, relationship to affected children, days per week of caregiving responsibilities, education level) about participant completing survey.

In total, the survey should take no more than 15 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Family members, specifically a parent, legal guardian, or relative, of a child who meets the following:

   * Age 3 to 17 years old at the time of survey completion
   * Reported diagnosis of a PTEN mutation
2. Enrollment in the RDCRN Contact Registry

Exclusion Criteria:

1. Inability to provide informed consent and complete survey
2. Inability to read and understand English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Families of children with PTEN mutation that are enrolled in the RDCRN Contact Registry.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Online Survey completed by family member(s) of affected child(ren) with PTEN | 3 months
  The survey will collect information regarding number of affected children in household, PTEN mutation type of effected children, age and gender of effected children, Age, neurodevelopmental disorders, medical problems, IQ, and access to clinical care (specialists currently being seen, specialists not able to see and why) of most affected child, research methods and mediums for disorder-specific treatment options for affected children, reasons behind not participating in clinical research options, and Facts (gender, age, if PTEN mutation carrier, work status, relationship to affected children, days per week of caregiving responsibilities, education level) about participant completing survey.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] Frazier TW, Embacher R, Tilot AK, Koenig K, Mester J, Eng C. Molecular and phenotypic abnormalities in individuals with germline heterozygous PTEN mutations and autism. Mol Psychiatry. 2015 Sep;20(9):1132-8. doi: 10.1038/mp.2014.125. Epub 2014 Oct 7. PMID 25288137
- [Background] Yehia L, Eng C. PTEN Hamartoma Tumor Syndrome. 2001 Nov 29 [updated 2025 Aug 7]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1488/ PMID 20301661
- [Background] Hansen-Kiss E, Beinkampen S, Adler B, Frazier T, Prior T, Erdman S, Eng C, Herman G. A retrospective chart review of the features of PTEN hamartoma tumour syndrome in children. J Med Genet. 2017 Jul;54(7):471-478. doi: 10.1136/jmedgenet-2016-104484. Epub 2017 May 19. PMID 28526761
- [Background] Nelen MR, Kremer H, Konings IB, Schoute F, van Essen AJ, Koch R, Woods CG, Fryns JP, Hamel B, Hoefsloot LH, Peeters EA, Padberg GW. Novel PTEN mutations in patients with Cowden disease: absence of clear genotype-phenotype correlations. Eur J Hum Genet. 1999 Apr;7(3):267-73. doi: 10.1038/sj.ejhg.5200289. PMID 10234502
- [Background] Pilarski R. Cowden syndrome: a critical review of the clinical literature. J Genet Couns. 2009 Feb;18(1):13-27. doi: 10.1007/s10897-008-9187-7. Epub 2008 Oct 30. PMID 18972196